CLINICAL TRIAL: NCT00005396
Title: Motivating Smokers--Reduce Child Environmental Tobacco Smoke Exposure
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4304; R01HL054351 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2002-04

CONDITIONS: Lung Diseases
MeSH Terms: conditions — Lung Diseases

SUMMARY:
To evaluate the efficacy of a motivational intervention designed to reduce children's exposure to environmental tobacco smoke in the household and to increase parental motivation towards smoking cessation.

DETAILED DESCRIPTION:
BACKGROUND:

The study tested the hypothesis that motivational intervention would yield greater reduction in smoking-related indices, compared to a usual care comparison condition. The study also predicted that the motivational intervention would differentially impact on cognitive and behavioral mediating mechanisms that accelerate behavior change and maintenance. Finally, the study tested the hypothesis that the motivational intervention would yield greater reduction in household exposure to environmental tobacco smoke (ETS), and therefore would also result in a significantly reduced number of children's respiratory illnesses.

DESIGN NARRATIVE:

This study utilized a community health center that served a low SES population in Rhode Island. The population was approximately 40 percent Hispanic and 45 percent Caucasian. Subjects were randomized to two intervention conditions:(1) a motivational intervention, that utilized self-help, telephone counselor calls, and motivational interviewing to provide feedback about children's health status and household concentrations of nicotine; (2) usual care, which included provision of self-help materials only. A repeated measures design was used (baseline, 3- and 6-month follow-ups). Outcome measures included household nicotine concentrations, movement through the stages of readiness to change, smoking cessation attempts, point-prevalence abstinence rates, and children's health status.

Several important public health priorities for research in lung health and prevention were targeted in this study, including: (1) reduction of ETS exposure among children from low income families, a group that has had a particularly high prevalence of chronic ETS exposure;. (2) development and evaluation of an intervention that was specifically tailored to match the characteristics of smokers who were low in motivation to quit smoking, a group that constituted 80 percent of the lower SES smoking population, yet that had been largely ignored in smoking research; (3) smoking intervention with an underserved, low-income and ethnic population that had poor access to standard approaches to smoking cessation and a particularly high smoking prevalence (household smoking prevalence = 60 percent); and (4) assessment of the impact of reductions in household ETS exposure on the respiratory health of children in the context of a longitudinal study.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1994-09; Study Completion 1999-08 (Actual)

REFERENCES:
- [Background] Emmons KM, Hammond SK, Fava JL, Velicer WF, Evans JL, Monroe AD. A randomized trial to reduce passive smoke exposure in low-income households with young children. Pediatrics. 2001 Jul;108(1):18-24. doi: 10.1542/peds.108.1.18. PMID 11433049